CLINICAL TRIAL: NCT06800508
Title: Comparison of Primary and Secondary Stability of a One-Piece Compressive Conometric Implant System in a Posterior Upper and Lower Jaw Clinical Study
Brief Title: Primary and Secondary Stability of a One-Piece Compressive Implant System
Status: Recruiting | Type: Observational
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Sarhang Gul, Principal investigator, University of Sulaimani
Other Study IDs: 227/24
Record Dates: First submitted 2025-01-17; First posted 2025-01-30 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Dental Implant
Keywords: Dental implant; primary stability; secondary stability; Compressive Implant; Conometric; One-piece implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One-piece implant: Preoperative CBCT for the implant area will be taken for analysis of anatomical features for all patients. Elastomeric impression will be obtained of both maxillary and mandibular arches, laboratory stone study casts will be made, and acrylic with metal sleeve surgical guide will be fabricated to localize the implant insertion position in the jaw bone without flap.
  After the administration of infiltration local anesthesia, the surgical guide will be fixed in its position on the jaw arch, and a drilling sequence will be applied according to the manufacturer's instructions to create a hole for implant placement. The compressive one-piece implant (fixture and abutment) from ROOTT Trade Company will be inserted with appropriate neck and abutment length. The implant insertion torque will be adjusted to 35 Ncm by the wrench.

SUMMARY:
Implant stability plays a major role in establishing implant osseointegration; it is considered an important requirement to decide the functional loading time with a fixed prosthesis. Objectives: to investigate the influence of one-piece implant position on their primary and secondary stability. The implant gains its Primary stability at placement time as a mechanical phenomenon that is related to the type of implant, placement technique used, and the local bone quality and quantity whereas, secondary stability is attributable to bone formation at the implant/tissue interface and in the surrounding bone. This study compares the stability of a compressive Conometric implant designed by Trade Company (ROOTT compressive with Conometric) in the posterior upper and lower jaws and optimizes the time of functional loading. This study's hypothesis is that implant stability is unaffected by the implant's position within the mouth cavity.

DETAILED DESCRIPTION:
Although Implant stability plays a major role in establishing the implant osseointegration, it is considered an important requirement to decide the functional loading time with a fixed prosthesis. Controlled loading is beneficial to maintain the implant stability during the early stage of healing as determined by resonance frequency analysis (RFA) measurement. There are different methods to determine implant stability, clinically examining the mobility by manual instrument, insertion torque value (ITV), electronic instrument, and radiograph evaluation of the bone around the implant; researchers found these are not sensitive enough. The introduction of quantitative methods, including the use of an RFA device (Osstell ISO, Integration Diagnostics AB, Gothenburg, Sweden) to measure implant stability, can yield valuable information, and its value range100. In contrast, a value greater than 70 is considered to indicate higher implant stability. Damping Capacity Analysis (DCA) device (Periotest; Medizintectechnik Gulden, Modautal, Germany) is another noninvasive method introduced to measure implant stability. Recently, Anycheck ( Neobiotech Seoul, Korea) is a modified DCA device introduced to measure implant stability, and Its value ranges from 1 to 99. Implant stability values of 1-59 were considered low stability; values of 60-64 indicated moderate stability; and values above 65 indicated high stability. The implant gains its Primary stability at placement time as a mechanical phenomenon that is related to the type of implant, placement technique used, and the local bone quality and quantity whereas, secondary stability is attributable to bone formation at the implant/tissue interface and in the surrounding bone. evaluated two-implant system stability using Periotest four months after the implant placement showed a mean of -1.9 for system A and mean of -2.1 system B whereas, Negative readings denote higher stiffness and a higher degree of osseointegration which indicated that implants were well osseointegrated and stable. Searching literature shows that applying different approaches to immediate loading can lead to survival rates in controlled studies comparable with those of conventionally loaded implants- however, this study is based on a small number. The selection of implant retained prosthesis type is a challenge for the dentist. Commonly there are different types of prosthesis retained to fixtures such as removable with precision attachment to the fixture and fixed restoration retained to the fixture either with cement or screw. Both cement and screw-retained fixtures have advantages and disadvantages like loos screw from time to time and remnant of cement under the restoration that leads to ridge mucous trauma. Conometric is another method to achieve retention of the prosthesis to the implant abutment, in addition to conventional cement and screw-based methods. Conometric works on the principle of frictional contact and elastic deformation of the connecting coping. Morse taper Conometric system used as implant-supported fixed dental prostheses retention found that the taper Conometric system can provide a retentive performance between implants and dental prostheses if proper insertion force is applied compared with cemented type without compromising the mechanical functionality of the system. Introduction One-piece implants with compressive threads, by ROOTT Implant Company, can be used for multiple units' restoration with immediate loading when adequate bone tissue is available. Studying the stability of a one-piece and comparing it to a two-piece implant suggested that both implant systems are clinically successful for dental rehabilitation and give consistent, longstanding results. Recently, this compressive implant was introduced with Conometric titanium caps (TEC) of different sizes and lengths. This study was conducted to compare the stability of a compressive Conometric implant designed by Trade Company (ROOTT compressive with Conometric) in the posterior upper and lower jaws and optimize the time of functional loading. This study's hypothesis is that implant stability is unaffected by the implant's position within the mouth cavity.

ELIGIBILITY:
Inclusion Criteria:

1. participating in this study already they are visiting the practice seeking implants to replace their missing teeth.
2. All teeth that want to be replaced with an implant should be extracted for more than two months.
3. Having enough height and width of alveolar bone to allow dental implant placement.

Exclusion Criteria:

1. Patients with systemic disease that could promise osseointegration.
2. Patients received radiation therapy in the head and neck region within the previous 12 months.
3. Smoker more than 10 cigarettes per day.
4. pregnant or lactating.
5. previous treatment with bisphosphonates.
6. presence of active periodontics infection.

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects seeking dental implant for missing teeth.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary dental implant stability | immediately after dental implant insertion as base line then at 3 and 6 month.
  Dental implant stability will be measured by resonance frequency analysis.

SECONDARY OUTCOMES:
Secondary dental implant stability | 3 and 6 months after dental implant insertion.
  Dental implant stability will be measured by resonance frequency analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sarhang S Gul, PhD, Principal Investigator — University of Sulaimani
Locations (1):
- A to Z dental care center, Sulaymaniyah, Iraq

IPD SHARING:
Plan to Share IPD: No
Only anonymous data about the participants will be reported in the study.

REFERENCES:
- [Result] Claudino D, Traebert J. Malocclusion, dental aesthetic self-perception and quality of life in a 18 to 21 year-old population: A cross section study. BMC Oral Health. 2013;13:2-7. https://doi.org/10.1186/1472-6831-13-3 Ali MA, Yassir YA. Mandibular Clinical Arch Forms in Iraqi Population: A National Survey. Diagnostics. 2022;12:1-15. https://doi.org/10.3390/diagnostics12102352 Najm AA, Mahdi AS, Al-Sudani RJ. Prevalence of Dental Anomalies among Iraqi Dental Students. J Baghdad Coll Dent. 2016;28:72-6. https://doi.org/10.12816/0033214 Moreno Uribe LM, Miller SF. Genetics of the dentofacial variation in human malocclusion. Orthod Craniofacial Res. 2015;18:91-9. https://doi.org/10.1111/ocr.12083 Staudt CB, Kiliaridis S. Different skeletal types underlying Class III malocclusion in a random population. Am J Orthod Dentofac Orthop. 2009;136:715-21. https://doi.org/10.1016/j.ajodo.2007.10.061 Abdulhussein ZA, Aksoy A. Compliance of Patients with Class III Malocclusion to Orthodontic Treatment. J Baghdad Coll Dent. 2022;34:12-24. https://doi.org/10.26477/jbcd.v34i1.3087 Mossey PA. The heritability of malocclusion: Part 1--Genetics, principles and terminology. Br J Orthod. 1999;26:103-13. https://doi.org/10.1093/ortho/26.2.103 Xue F, Wong RWK, Rabie ABM. Genes, genetics, and Class III malocclusion. Orthod Craniofacial Res. 2010;13:69-74. https://doi.org/10.1111/j.1601-6343.2010.01485.x Hussein AS, Porntaveetus T, Abid M. The association of polymorphisms in BMP2/MYO1H and skeletal Class II div.1 maxillary and mandibular dimensions. A preliminary 'report. Saudi J Biol Sci. 2022;29:1-7. https://doi.org/10.1016/j.sjbs.2022.103405 Manolio TA. Genomewide Association Studies and Assessment of the Risk of Disease. N Engl J Med. 2010;363:166-76. https://doi.org/10.1056/NEJMra0905980 Weiler CA, Drumm ML. Genetic influences on cystic fibrosis lung disease severity. Front Pharmacol. 2013;4:1-19. https://doi.org/10.3389/fphar.2013.00040 Strauss JF, Romero R, Gomez-Lopez N, Haymond-Thornburg H, Modi BP, Teves ME, et al. Spontaneous Preterm Birth: Advances toward the Discovery of Genetic Predisposition. Am J Obstet Gynecol. 2018;218:294-314. https://doi.org/10.1016/j.ajog.2017.12.009 Weaver CA. Candidate Gene Analysis of 3D Dental Phenotypes in Patients with Malocclusion. University of Iowa; 2014. Little J, Higgins JPT, Ioannidis JPA, Moher D, Gagnon F, Elm EV, et al. STrengthening the REporting of genetic association studies (STREGA)- An extension of the STROBE statement. Genet Epidemiol. 2009;33:581-98. https://doi.org/10.1002/gepi.20410 Steiner CC. Cephalometrics for you and me. Am J Orthod. 1953;39:729-55. https://doi.org/10.1016/0002-9416(53)90082-7 Guo L, Feng Y, Guo HG, Liu BW, Zhang Y. Consequences of orthodontic treatment in malocclusion patients: Clinical and microbial effects in adults and children. BMC Oral Health. 2016;16:1-7. https://doi.org/10.1186/s12903-016-0308-7